CLINICAL TRIAL: NCT06486636
Title: Pericardiotomy in Cardiac Surgery Trial
Brief Title: Pericardiotomy in Cardiac Surgery
Acronym: PRINCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: McMaster University (Other); Hamilton Health Sciences Corporation (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRINCE - 2024
Record Dates: First submitted 2024-06-13; First posted 2024-07-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Cardiac Events
Keywords: Pericardiotomy; Cardiac Surgery; Hospital Readmission; Post-Operative Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Each patient will be assigned in a blinded fashion to one of two groups (left posterior pericardiotomy or no posterior pericardiotomy) in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding to allocation will be maintained for all parties, excluding the operating surgeon and necessary operating room personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left Posterior Pericardiotomy Group (Experimental): The surgeon will perform a left posterior pericardiotomy during the patient's cardiac surgery.
  Interventions: Procedure: Left Posterior Pericardiotomy
- No Posterior Pericardiotomy Group (No Intervention): The surgeon will not perform a posterior pericardiotomy during the patient's cardiac surgery.

INTERVENTIONS:
Procedure: Left Posterior Pericardiotomy — The surgeon will perform a left posterior pericardiotomy while the patient is on cardiopulmonary bypass. A soft channel drain will be put into place at an angle directed toward the posterior pericardium. The surgeon will grasp the pericardium and use cautery to make a 4- to 5-cm opening between the left inferior pulmonary vein and the diaphragm. The previously prepared channel drain is cut to the desired length and placed through the pericardiotomy along the diaphragm and into the pleural space.
  Arms: Left Posterior Pericardiotomy Group

SUMMARY:
PRINCE is an international, multicentre, randomized controlled trial of posterior pericardiotomy in patients without a history of atrial fibrillation (AF) or flutter undergoing cardiac surgery.

DETAILED DESCRIPTION:
Approximately 30% of cardiac surgical patients develop post-operative atrial fibrillation (POAF). Its incidence varies depending on the type of cardiac operation. POAF is associated with short- and long-term adverse events, including mortality, stroke, and heart failure. POAF has also been significantly associated with unplanned hospitalization for heart failure.

During cardiac surgery, pericardial fluid tends to collect posterior to the left atrium. Even small amounts of fluid may trigger atrial arrhythmias. A posterior left pericardiotomy is a surgical procedure that involves cauterizing an opening between the left inferior pulmonary vein and the diaphragm. This procedure may allow for more prolonged drainage of the pericardial fluid into the left pleural space. Recent research evidence found that posterior pericardiotomy was associated with a significantly lower incidence of POAF.

The existing data on posterior pericardiotomy is promising for a reduction in POAF. However, no high-quality study has demonstrated that this reduction improves clinical outcomes in the years after cardiac surgery. The PRINCE trial's long-term follow-up of patients randomized to left posterior pericardiotomy could conclusively demonstrate whether the relationship of POAF to post-discharge clinical outcomes is causal and modifiable.

The PRINCE trial will evaluate the effectiveness and safety of posterior left pericardiotomy in preventing POAF and improving post-discharge clinical outcomes in a broad spectrum of cardiac surgery patients.

The intervention under investigation is left posterior pericardiotomy which is compared to no posterior pericardiotomy during cardiac surgery. The early co-primary outcome is in-hospital POAF, and the late co-primary outcome is the hierarchical composite of time to all-cause death, time to ischemic stroke, time to systemic arterial embolism, time to unplanned hospital visit/readmission for cardiac reasons, and time to atrial fibrillation after index hospital discharge.

The study will enrol 1400 patients from 30 centres, globally. Follow-up visits will be performed in person or by telephone 1 and 6 months post-randomization (+7 days), and then every 6 months (+30 days) until an average follow-up of 5 years for the study participants (estimated to be 4 years after completion of enrolment).

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years of age
* Requiring surgical intervention on the proximal aorta, cardiac valves, and/or coronary arteries
* Able to provide informed consent

Exclusion Criteria:

* History of atrial fibrillation or flutter
* Cardiac surgery procedures not included in the inclusion criteria (planned ventricular assistance device, aortic arch, transplantation surgery)
* Prior cardiac surgery requiring opening of the pericardium
* Previous surgical instrumentation of the left pleural cavity
* Patient undergoing minimally invasive cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital post-operative atrial fibrillation | Within 5 days after index cardiac surgery
  Number of patients with post-operative atrial fibrillation within the first 5 days postoperatively or up to hospital discharge, whichever occurs first
Hierarchical composite of all-cause death, ischemic stroke, systemic arterial embolism, unplanned hospital visit/readmission for cardiac reasons, and atrial fibrillation. | Over the duration of the follow-up period to a common end date (mean follow-up of 5 years).
  Number of patients with a composite of all-cause death, ischemic stroke, systemic arterial embolism, unplanned hospital visit/readmission for cardiac reasons, and atrial fibrillation events, evaluated using the win ratio (thereby accounting for the difference in importance of these outcomes).

SECONDARY OUTCOMES:
Post-operative atrial fibrillation (POAF) | Over the duration of the follow-up period to a common end date (mean follow-up of 5 years).
  Number of patients with post-operative atrial fibrillation
Length of post-operative in-hospital stay | Over the duration of the follow-up period to a common end date (mean follow-up of 5 years).
  Length of time the patient in hospital after their index cardiac surgery
Pericardial effusion without tamponade | From index surgery completion to within 30 days of index surgery
  Number of pericardial effusions that occur, excluding cardiac tamponade
Death | From index surgery completion to within 30 days of index surgery
  Occurrence of death
Ischemic stroke or systemic arterial embolism | From index surgery completion to within 30 days of index surgery
  Number of ischemic strokes or systemic arterial embolisms
Hospital readmission or unplanned hospital visit | From index surgery completion to within 30 days of index surgery
  Number of hospital readmissions or unplanned hospital visits
Quality of life assessed by the European quality of life index version 5D (EQ-5D-5L) questionnaire | Over the duration of the follow-up (mean follow-up of 5 years)
  The EQ-5D-5L consists of a descriptive system and the EQ visual analogue scale (EQ VAS) scale of 0-100 where the endpoints are labelled 'The best health you can image' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is measured on a 5 point scale: no problems, slight problems, moderate problems, severe problems and extreme problems.

OTHER OUTCOMES:
Number of patients with phrenic nerve injuries | Within 30 days of index surgery
  Safety outcome
Number of patients with left pleural interventions | Within 30 days of index surgery
  Safety outcome
Number of patients with esophageal injuries | Within 30 days of index surgery
  Safety outcome
Number of patients requiring re-operation for bleeding | Within 48 hours of index surgery completion
  Safety outcome
Number of patients with cardiac tamponade | Within 30 days of index surgery
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, Principal Investigator — Population Health Research Institute; Emilie Belley-Côté, Principal Investigator — Population Health Research Institute; Mario Gaudino, Principal Investigator — Weill Medical College of Cornell University; Sigrid Sandner, Principal Investigator — Medical University Vienna; Björn Redfors, Principal Investigator — Göteborg University
Locations (4):
- Weill Cornell Medicine, New York, New York, United States
- Medical University Vienna, Vienna, Vienna, Austria
- Hamilton Health Sciences, Hamilton, Ontario, Canada
- University of Foggia, Policlinico Foggia, Foggia, Foggia, Italy